CLINICAL TRIAL: NCT01694693
Title: Description of Joint Population and Assessment of Impact on Health Status of Orencia in Patients With Rheumatoid Arthritis in France. A Database Analysis Based on SFR's ORA Long-term Cohort Study
Status: Withdrawn | Type: Observational
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-364
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients treated by Orencia: RA patients treated by Orencia according to usual practice from June 1st 2007
  Interventions: Drug: Orencia

INTERVENTIONS:
Drug: Orencia — No Intervention

SUMMARY:
Database analysis:

* To describe how Orencia is prescribed in France in Rheumatoid Arthritis (RA)
* To describe joint population of Orencia
* To assess the impact of the treatment on health status of the treated population as assessed by morbid-mortality criteria
* To describe therapeutic strategies and use of health services

DETAILED DESCRIPTION:
* Observational Model: Historic cohort generated from Société Française de Rhumatologie's (SFR) Orencia and Rheumatoid Arthritis (ORA) registry
* Sampling Method: all physicians and sites taking in charge RA patients received an invitation mailing to participate to ORA
* Minimum Age: 18 years old at Orencia initiation

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Adult outpatients, male or female aged ≥ 18 years old
* Diagnosed with a rheumatoid arthritis according to ACR criteria
* Treated with Orencia according to usual practice conditions from June 1st 2007
* Agreeing to participate

Exclusion Criteria:

* Patients treated by Orencia in the context of clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in SFR's ORA Registry
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01-31 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with first clinically significant Disease Activity Score (DAS) change | Up to 5 Years
  Change from DAS28 [C - reactive protein (CRP) and erythrocyte sedimentation rate (ESR)] measured at treatment initiation ≥ 1.2
  DAS28 will be measured every 6 months during 5 years
Number of patients with first response to treatment [according to definition of European League Against Rheumatism (EULAR) response criteria] | Up to 5 Years
  EULAR response will be measured every 6 months during 5 years
Number of patients with first Low Disease Activity State (LDAS) | Up to 5 Years
  Change from DAS28 [C - reactive protein (CRP) and erythrocyte sedimentation rate (ESR)] measured at treatment initiation ≤ 3.2
  DAS28 will be measured every 6 months during 5 years
Number of patients with first Remission state | Up to 5 Years
  Change from DAS28 [C - reactive protein (CRP) and erythrocyte sedimentation rate (ESR)] measured at treatment initiation <2.6
  DAS28 will be measured every 6 months during 5 years
Number of patients disease progression with prior improvement | Up to 5 Years
Number of patients disease progression with no prior improvement | Up to 5 Years
Number of patients with modification of Orencia administration condition | Up to 5 Years
Number of patients discontinued and switched from Orencia | Up to 5 Years
Incidence rate of any type of Adverse events related to Orencia | Up to 5 Years
Number of patients with specific predefined events | Up to 5 Years
  Predefined events are severe infection, thromboembolic events, cancer, lymphoma, other autoimmune disease, cutaneous disorder, significant or persistent disability, death
Response over the time will be assessed over 5 years on EULAR response, LDAS | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx